CLINICAL TRIAL: NCT05452967
Title: Comparison of Pain Scores by Using Audiovisual Distraction Aids in Post Operative Paediatric Patients.
Brief Title: Comparison of Pain Scores by Using Audiovisual Aids.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Shemila Abbasi, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2172-14474
Record Dates: First submitted 2021-12-09; First posted 2022-07-12 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2022-07

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Group C (conventional analgesia group) Group CD (conventional analgesia plus distraction technique)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional analgesia group Group C (No Intervention): this group will receive rescue analgesia as per need
- Distraction group: Group CD (Experimental): This group will be distracted with the help of mobile or tablet and then will assess that rescue analgesia will be needed in post anaesthesia care unit or not
  Interventions: Other: Distraction technique

INTERVENTIONS:
Other: Distraction technique — The post operative pediatric patients will be given mobile phone in recovery for plying games and watching cartoons and with the help of this distraction technique will assess that routine rescue analgesia is needed or not
  Arms: Distraction group: Group CD

SUMMARY:
This study will be conducted at post anaesthesia care unit of Department of Anesthesiology, Aga Khan University Hospital Karachi.

The aim of this study is to compare the post operative analgesia between two groups of post operative paediatric patients, Conventional group, receiving conventional analgesia and the group of patients in which distraction technique will be used. Conventional group will only receive conventional analgesia while the distraction group will receive conventional analgesia as well as distraction technique. Distraction technique that will be used is a non-pharmacological method of pain relief for post-operative paediatric patients in post anesthesia care unit. (games on tablets, listening poems, watching cartoons). Conventional analgesia is the standardise rescue analgesia of intravenous administration of analgesics in post anaesthesia care unit prescribed. The analgesia will include I/V Tramadol 0.5 to 1mg/kg and Paracetamol 10mg/kg).

Our primary outcome will be pain scores using Wong-Baker FACES® pain rating scale and parent's satisfaction as secondary outcome.

DETAILED DESCRIPTION:
The main purpose of this study is to compare the post operative analgesia between two groups (Conventional and the Distraction Group ) receiving conventional analgesia with or without distraction technique. Conventional group will only receive conventional analgesia while group Distraction group will receive conventional analgesia as well as distraction technique.

This randomised controlled trial will be conducted at post anaesthesia care unit of Department of Anesthesiology, Aga Khan University Hospital Karachi after approval by Ethical Review committee. After getting registration from clinical trials, the data will be collected. The purpose along with procedure of the study will be explained to the parents/guardian and informed consent will be taken in the ward. Patients will be divided into two equal groups by computer generated random number and the information will be provided to the investigator in the form of sealed envelopes which will not be opened until patient consent is obtained. The information and the demographics of the patients will be entered in the proforma attached as annexure. Data will be collected in the pre designed form. For the purpose of data collection the form is divided into two sections: SECTION I: - This section will be filled by the primary investigator in operation room. SECTION II: - This section will be completed by the data collector in PACU.

When the investigator will receive patients in post anaesthesia care unit, the nurse will be informed about the allocated group. Parents will be present with both groups. Patients in the conventional group will receive their routine rescue analgesics. While patients in the group distraction group will be engaged in distraction methods once the child is awake and his/her response will be noted in form II at given intervals by data collector. Heart Rate, Blood pressure, oxygen saturation and respiratory rate will be noted from the monitors. The pain score will be noted with the help of given Wong Baker faces pain scale (The first face represents a pain score of 0, and indicates "no hurt". The second face represents a pain score of 2, and indicates "hurts a little bit." The third face represents a pain score of 4, and indicates "hurts a little more". The fourth face represents a pain score of 6, and indicates "hurts even more"). on proforma. Routine rescue analgesia (Injection Paracetamol; 15 mg/Kg and Injection Nalbuphine 1/4 dose of the intra operative dose) will be used if patient still experiences pain. The study will be concluded at discharge from the post anaesthesia care unit. These children will be given tablets/smart phone to choose one of the options like playing games, to listening poems and watching cartoons.

It will be the responsibility of primary investigator with assistance of data collector. Primary investigator will ensure the study protocol compliance. A copy of the consent form taken will be attached with proforma. The confidentiality of the patient and data will be maintained by assigning a number for each patient data. The electronic data will be password protected and hard copies will be kept in research cell in locked cupboard.

At the completion of the study, results will be shared with the parents upon their request. Public disclosure includes publication of an abstract or full paper in a scientific journal and presentation at a scientific meeting.

ELIGIBILITY:
Inclusion Criteria:

1. All elective cases on pediatric lists including Orthopaedics, plastic surgery, paediatrics surgery.
2. ASA level I and II with age range between 3 and 7 years will be included in the study.

Exclusion Criteria:

1. All pediatric patients who are neurologically challenged,
2. Undergoing head and neck surgery,
3. Patients undergoing emergency surgery,
4. cases with difficult airway,
5. language barrier and whose parents have not consented to participate in the study will be excluded.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of pain scores by using audiovisual distraction aids in post operative paediatric patients. | Baseline data (hemodynamic variables and pain score) on arrival in the post anaesthesia care unit . First reading at 15 minutes after intervention. Second at 30 minutes and last at 45 minutes. All the readings will be compared with the initial baseline.
  The pain scores will be assessed in post anaesthesia care unit by using Wong Baker FACES pain rating scale. This scale comprises of a series of faces ranging from a happy face at "0" or "no hurt" to a crying face at "10" which represents the worst pain imaginable. The higher the score the worse will be the pain. We will use a proforma for data collection and for measuring the desired outcome.

SECONDARY OUTCOMES:
Comparison of pain scores by using audiovisual distraction aids in post operative paediatric patients. | After concluding /last reading at 45 minutes parents satisfaction will be assessed.
  Parent's satisfaction will be assessed once the patient will be signed off from the post anaesthesia care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Shemila Abbasi, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT05452967/Prot_000.pdf
  • Informed Consent Form (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT05452967/ICF_001.pdf